CLINICAL TRIAL: NCT04442087
Title: Seroprevalence of Anti-SARS-CoV2 Among Children According to Parents' SARS-CoV2 Serological Status. Study in a Hospital Population Assistance Publique-Hôpitaux Paris
Brief Title: Study of Seroprevalence of Anti-SARS-CoV2 Among Children of Hospital Workers in AP-HP
Acronym: FamilyPEDCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200627; 2020-A01480-39 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-06-08; First posted 2020-06-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: SARS-CoV2
Keywords: SARS-CoV2; COVID-19; Serology; Hospital workers; Children
MeSH Terms: conditions — COVID-19 | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Serology SARS-CoV2 — Collect serum for Serology SARS-CoV2 at inclusion
Behavioral: Data collection — Collect clinical and demographic data, habitus, Lifestyle Counseling at inclusion

SUMMARY:
The purpose of this study is to define seroprevalence of anti-SARS-CoV2 among children of Hospital Workers in APHP, particularly exposed population, according to parents' SARS-CoV2 serological status.

ELIGIBILITY:
Inclusion Criteria:

Hospital workers :

1. Individuals aged over 18, having a professional activity at the APHP (employees, interns, volunteers)
2. Affiliated to a social security regimen
3. Have at least one child under the age of 18 living in the same house.
4. have signed consent

Child (ren), spouse and other member (s) residing at household:

Child (ren), spouse and any other member residing in the household of a professional of the Paris Center Hospitals meeting the inclusion criteria above.

Exclusion Criteria:

Refuse to participate in research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of antibodies anti- SARS Cov2 in blood sample of children of Hospital workers | at inclusion
  Percentage of children with seropositive in blood sample according to parents' SARS Cov2 serological status
Seroprevalence of antibodies anti- SARS Cov2 in saliva sample of children of Hospital workers | at inclusion
  Percentage of children with seropositive according in saliva sample to parents' SARS Cov2 serological status

SECONDARY OUTCOMES:
Number of Asymptomatic Children with a positive seroloy | At inclusion
Number of severely symptomatic Children with a positive serology | At inclusion
Prevalence of different clinical symptoms in children with a positive serology | At inclusion
Serological result of each member of the family | At inclusion
Number of spouses of hospital workers with a positive serology | At inclusion
Number of Asymptomatic spouses of hospital workers with a positive serology | At inclusion
Number of severely symptomatic spouses of hospital workers with a positive serology | At inclusion
Comparison of Serological result obtained in blood and saliva samples | At inclusion
Risk factors based on a questionnaire for children and adults | At inclusion
  the following factors will be of particular importance: characteristics and composition of the family home, barrier measures, medical history and comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Solen KERNEIS, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Flore ROZENBERG, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Jean-Marc TRELUYER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre d'investigation clinique (CIC) Necker Cochin in Necker Children's Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No